CLINICAL TRIAL: NCT01377558
Title: Effects of Different Types of Exercise Interventions in Patients With Type 2 Diabetes - Aerobic Endurance Training Versus Strength Endurance Training Versus Combined Aerobic Endurance and Strength Endurance Training -
Brief Title: Effects of Different Types of Exercise Interventions in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Giessen (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Andree Hillebrecht, Dr. med., Department of Sports Medicine Giessen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gi-03-2011
Record Dates: First submitted 2011-06-09; First posted 2011-06-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes
Keywords: aerobic training; resistance training; combination of aerobic and resistance training; diabetes; type 2 diabetes; HbA1c; endothelial dysfunction; inflammation markers; Parodontitis; Exercise intervention; training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Dry Socket

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aerobic endurance training intervention (Experimental): Aerobic endurance training
  Interventions: Other: Aerobic endurance training intervention
- Strength endurance training intervention (Experimental): Strength endurance training
  Interventions: Other: Strength endurance training intervention
- Combined training intervention (Experimental): Combined aerobic endurance training and strength endurance training intervention
  Interventions: Other: Combined aerobic endurance and strength endurance training
- Control group (No Intervention): control group

INTERVENTIONS:
Other: Aerobic endurance training intervention — The aerobic endurance training group will use cardiovascular training devices
  week 1-4: 15 minutes warm up (group) 15 minutes intervention at 80-100% vAT two times per week
  week 5-13: 15 minutes warm up (group) 30 minutes intervention at 95-110% vAT two times per week
  week 14-26: 15 minutes warm up (group) 45 minutes intervention at 95-110% vAT two times per week
  Other Names: aerobic endurance training
  Arms: Aerobic endurance training intervention
Other: Strength endurance training intervention — The strength endurance training intervention group will perform eight exercises on weight machines (Milon circuit training- 60 seconds activity, 30 seconds break)
  week 1-4: 15 minutes warm up (group) 1 session resistance training intensity 3 (Buskies) two times per week
  week 5-13: 15 minutes warm up (group) 2 sessions resistance training intensity 5 (Buskies) two times per week
  week 14-26: 15 minutes warm up (group) 3 sessions resistance training intensity 5 (Buskies) two times per week
  Other Names: Strength endurance training
  Arms: Strength endurance training intervention
Other: Combined aerobic endurance and strength endurance training — week 1-4: 15 minutes warm up (group) 15 minutes intervention at 80-100% vAT once per week and 15 minutes warm up (group) 1 session resistance training intensity 3 (Buskies) once per week
  week 5-13: 15 minutes warm up (group) 15 minutes intervention at 95-110% vAT and 1 session resistance training intensity 5 (Buskies) two times per week
  week 14-26: 15 minutes warm up (group) 30 minutes intervention at 95-110% vAT and 1 session resistance training intensity 5 (Buskies) once a week and 15 minutes warm up (group) 15 minutes intervention at 95-110% vAT and 2 sessions resistance training intensity 5 (Buskies) once a week
  Arms: Combined training intervention

SUMMARY:
The purposes of the study are

* to determine which kind of supervised exercise intervention (aerobic endurance training versus strength endurance training versus combined aerobic endurance and strength endurance training) is more effective in improving the metabolic parameters in typ 2 diabetes patients
* to investigate what kind of intervention is more successful in reduction of concomitant diseases and improving quality of life
* to assess what kind of intervention induces highest effects in long term persistence of these positive changes

DETAILED DESCRIPTION:
Meta-analyses which evaluated the effects of structured exercise programs in patients with type 2 diabetes demonstrate that regular physical activity improves glycosylated haemoglobin (König et al.: Resistance Exercise and Type 2 Diabetes Mellitus, Deutsche Zeitschrift für Sportmedizin Jahrgang 62, Nr. 1 (2011): 5-9). Sigal et al. proved that either aerobic or resistance training alone improved glycemic control in type 2 diabetes, but the improvements are greatest with combined aerobic and resistance training (Sigal, RJ, et al.: Effects of Aerobic Training, Resistance Training, or Both on Glycemic Control in Type 2 Diabetes, Ann Intern Med. 2007 Sep 18;147(6):357-69).

Therefore, aim of the current study is to compare the effects of aerobic endurance training or resistance endurance training or the combination of aerobic endurance training and resistance endurance training in diabetes type 2 patients without any other lifestyle or dietary interventions.

ELIGIBILITY:
Inclusion Criteria:

* diagnoses of type 2 diabetes (ADA criteria)
* admitted diabetes treatments will be diet and oral hypoglycemic agents

Exclusion Criteria:

* sports intervention >60 minutes per week
* medical conditions
* preproliferative or proliferative retinopathy
* instable coronary heart disease
* inability to perform the scheduled physical activity programs
* acute clinically significant intercurrent diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c-level (haemoglobin A1c) | 6 months

SECONDARY OUTCOMES:
Change in HOMA-Index | 3 and 6 months
Change in beta-cell-function | 3 and 6 months
  Measured by OGTT (Oral Glucose Tolerance Test)
Change in fasting plasma glucose levels | 3 and 6 months
Change in total cholesterol levels | 3 and 6 months
Change in HDL-cholesterol levels | 3 and 6 months
Change in LDL-cholesterol levels | 3 and 6 months
Change in triglyceride levels | 3 and 6 months
Change in antidiabetic medications | 3 and 6 months
  Class and dosage of blood-glucose lowering drugs are recorded before, after 3 and 6 months
Change in inflammation markers | 3 and 6 months
  CrP, blood count, interleukinstatus, cytokinstatus
Change in body weight | 3 and 6 months
Change in body composition | 3 and 6 months
  by Bio-impedance analysis, waist to hip ratio, range of thigh
Change in strength | 3 and 6 months
  by Dr. Wolff Back Check
Change of maximum heart rate | 3 and 6 months
  Measured by an incremental exercise test
Change of peak oxygen uptake | 3 and 6 months
  Measured by an incremental exercise test
Change of vAT (ventilatory anaerobic threshold) | 3 and 6 months
  Measured by an incremental exercise test
Change in blood pressure | 3 and 6 months
Change in renal function | 3 and 6 months
  Creatininlevel, Albuminlevel (urine), Telomere length
Change in concentration | 3 and 6 months
  by d2-test
Change in quality of life | 3 and 6 months
  by questionnaire: SF-12, EQ5
Change of nutrition | 3 and 6 months
  by questionnaire: FEV, FFQ
Change in voluntary physical activity | 3 and 6 months
  meassured by pedometer (one week)
Change of cardiac output by Impedance cardiography | 3 and 6 months
  by Task Force Monitor
Change of barorezeptorsensitivity | 3 and 6 months
  by Task Force Monitor
Change in carotid-Intima-Media-Thickness | 3 and 6 months
Change in aortic pulse-wave velocity | 3 and 6 months
Change in central aortic pressure | 3 and 6 month
Change in endothelial dysfunction | 3 and 6 months
Change of parodontitis | 3 and 6 months
Follow up of all parameters mentioned above | after 12 months
  Follow up after 12 months (6 months after completing the exercise intervention) without any supervised intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andree Hillebrecht, Dr. med., Principal Investigator — University of Giessen
Locations (2):
- Germany (2):
  - University of Giessen, Giessen, Hesse
  - Sportpark Zwickau, Glauchau, Meerane, Zwickau, Saxony